CLINICAL TRIAL: NCT06129500
Title: CBT for Mood-Driven, Problematic, Impulsive Behaviours in Bipolar Disorder: A Case Series Evaluation
Brief Title: CBT for Problematic Impulsive Behaviours in Bipolar Disorder: A Case Series / CBT-PIB
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Paused due to change in staffing arrangements
Sponsor: University of Exeter (Other)
Collaborators: Southern Health NHS Foundation Trust (Other); Somerset NHS Foundation Trust (Other); Devon Partnership NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-23-07
Record Dates: First submitted 2023-10-26; First posted 2023-11-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Impulsivity; Bipolar Disorder; Hypomania; Bipolar I Disorder; Bipolar II Disorder; Bipolar Affective Disorder; Impulsive Behavior
MeSH Terms: conditions — Impulsive Behavior; Bipolar Disorder; Mania | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This project will follow an ABA case-series design.
  In an ABA design, for an individual receiving a treatment there is a measurement period (baseline) before the treatment phase, and then again after the treatment phase, to allow exploration of the apparent stability of any changes observed over the treatment period.
  Participants will be assigned to a two-week baseline phase, up to twelve-session intervention phase, and a two-week post-intervention phase. This will allow for three baseline measurements, to establish symptom and mood stability prior to treatment, and a two-week post-intervention measurement phase to explore the stability of any intervention-related changes.
  Symptoms will be measured weekly across the baseline period, treatment phase and post-treatment periods. Participants will also complete additional self-report measures and be invited to participate in a semi structured interview to gather qualitative feedback post treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT for mood driven, problematic, impulsive behaviours (Experimental): All participants will be offered the 12 week CBT intervention
  Interventions: Behavioral: Cognitive Behavioural Therapy for Problematic Impulsive Behaviours

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Problematic Impulsive Behaviours — Up to 12 sessions of Cognitive Behavioural Therapy adapted to focus on mood-driven impulsivity in adults with bipolar disorder.

SUMMARY:
The goal of this case series is to explore whether a talking therapy, specifically Cognitive Behavioural Therapy (CBT) is acceptable and feasible in the management of mood-driven impulsive behaviours in people with bipolar disorder (BD).

The main questions it aims to answer are:

* Whether CBT Is a feasible intervention for participants with BD who report mood-driven, problematic impulsive behaviours.
* Whether CBT for mood-driven, problematic impulsive behaviours (CBT-PIB) is acceptable to service users with BD and therapists.
* Whether clinical outcomes are consistent with the potential for this novel intervention to offer clinical benefit to participants with BD.

The study also hopes to:

* conduct a preliminary examination of the safety of CBT-PIB and the research procedures.
* gather information on the potential mechanisms of action of CBT-PIB and,
* gather information on the types of mood-driven impulsive behaviours individuals with BD may seek support for.

Participants will:

* be offered up to 12 individual sessions of CBT focusing on mood-driven impulsive behaviours.
* be asked to complete a battery of self-report measures (5) when they enter the study and at the start and end of treatment.
* be asked to track mood and impulsive behaviours by completing a brief set of measures (3) weekly during the two-week baseline phase, the intervention phase and the 2-week post-intervention phase.
* be asked to complete a survey on the acceptability of the intervention and
* be invited to an optional semi-structured interview on their research experience.

ELIGIBILITY:
Inclusion Criteria:

* meeting diagnostic criteria for Bipolar I or II Disorder (SCID-5- Structured clinical interview for depression )
* able to identify at least one impulsive, problematic behaviour to target during the intervention;
* participants will require working knowledge of written and spoken English, sufficient to be able to make use of therapy and to be able complete research assessments without the need of a translator.

Exclusion Criteria:

* major depressive episode (identified through SCID-DSM-5);
* current experience of mania;
* current/past learning disability (IQ of less than 70 with impairment of social and adaptive functioning)
* organic brain change or substance dependence (drugs and alcohol) that would compromise ability to use therapy;
* current marked risk to self (i.e. self-harm or suicide) that we deem could not be appropriately managed in by the therapy site;
* currently lacking capacity to give informed consent;
* currently receiving other psychosocial therapy for impulsivity or bipolar disorder;
* current engagement in another psychological intervention addressing bipolar disorder or impulsivity;
* presence of another area of difficulty that the therapist and client believe should be the primary focus of intervention (for example, Post-Traumatic Stress Disorder, psychosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2027-01-24 (Estimated)

PRIMARY OUTCOMES:
Overall acceptability and feasibility of the CBT protocol measured by the Client Satisfaction Questionnaire CBT-PIB | Post-intervention at week 16
  qualitative and quantitative feedback from participants
rates of clinically significant and reliable change in mood measured by the Patient health questionnaire (PHQ-9) | Through study completion, an average of 18 weeks
  used to monitor the severity of depression and response to treatment
rates of clinically significant and reliable change in symptoms of mania measured by the Altman Self-Rating Mania Scale | Through study completion, an average of 18 weeks
  scale that assesses the presence and severity of manic or hypomanic symptoms
Changes in management of impulsivity measured by the Visual Analogue Scale | Through study completion, an average of 18 weeks
  Visual scale measuring the severity and impact of general and behavioural impulsivity
Number of participants with intervention-related adverse events assessed by the adverse events form | Through study completion, an average of 18 weeks
  qualitative form eliciting adverse events

SECONDARY OUTCOMES:
rates of clinically significant and reliable change in general daily functioning as measured by the Work and Social Adjustment Scale | At baseline, 2 weeks and 14 weeks
  scale assesses changes in the impact of a person's mental health difficulties on their ability to function in terms of work, home management, social leisure, private leisure and personal or family relationships.
rates of clinically significant and reliable change in quality of life as measured by the Brief Quality of Life in Bipolar Disorder | At baseline, 2 weeks and 14 weeks
  self-report measure of changes in disorder-specific quality of life
rates of clinically significant and reliable change in symptoms of anxiety as measured by the General Anxiety Disorder Assessment (GAD7) | At baseline, in 2 weeks and in 14 weeks
  scale measuring changes in symptoms of anxiety
rates of clinically significant and reliable change in overall wellbeing as measured by the Warwick-Edinburgh Mental Well-being Scale | At baseline, in 2 weeks and in 14 weeks
  scale measuring changes in positive features of mental health
rates of clinically significant and reliable change in impulsivity measured by the Short Urgency, Premeditation (lack of), Perseverance (lack of), Sensation Seeking, Positive Urgency, Impulsive Behavior Scale | At baseline, in 2 weeks and in 14 weeks
  Scale measuring changes in 5 domains of impulsive behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Jan Freeman, MSc, Principal Investigator — University of Exeter
Locations (1):
- AccEPT Clinic, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All data that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Access will be possible from date of publication.
Access Criteria: The research database will be registered with the University of Exeter public access database. The dataset will be anonymous and will be registered with a metadata only record, allowing the research team to control access to the dataset, restricting it to appropriately qualified third parties.